CLINICAL TRIAL: NCT01192854
Title: A Multi-center, Randomized, Double-blind, Positive-control, Phase III Trial of the Efficacy and Safety of Clevudine
Brief Title: An Study of Efficacy and Safety of Clevudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XY3-III-CLV-1001A02.4
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Hepatitis B
Keywords: Clevudine; efficacy; safety; chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine; adefovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Clevudine
- 2 (Active Comparator)
  Interventions: Drug: Adefovir

INTERVENTIONS:
Drug: Clevudine — Clevudine flexible dosages of 30 mg/day
  Arms: 1
Drug: Adefovir — Adefovir flexible dosages of 10 mg/day
  Arms: 2

SUMMARY:
Randomized, double blind parallel group, positive control, multi-center trial. Patients will be randomized at 1:1 ratio in group A or group B

ELIGIBILITY:
1. Patients are between 18 and 65, inclusive.
2. All the male and female reproductive-aged subjects should use reliable and appropriate contraceptive method from the entrance of screening to at least 3 months within the end of study.
3. Hepatitis B virus Early Antigen (HBeAg) positive patient with HBV DNA >1 x 105 copies/ml, HBeAg negative patient with HBV DNA >1 x 104 copies/ml within 30 days of baseline.
4. Absolute neutrophil count > 1500 /mm3.
5. Alpha fetoprotein within normal laboratory limit at screening.
6. Normal electrocardiogram (ECG) or clinically non-significant changes at screening.
7. Able to participate and willing to give written informed consent before starting therapy.
8. Able and willing to comply with study assessments and restrictions.
9. Normal renal function to take Adefovir without any dose modifications; Creatinine clearance must be >50 ml/min (based on the Cockcroft-Gault equation.

Exclusion criteria

1. Subjects coinfected with human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV) or hepatitis E virus
2. Patients previously or currently treated with approved and investigational nucleosides (e.g.: lamivudine, adefovir. entecavir, lobucavir, famciclovir, tenofovir, telbivudine) for any duration.
3. Other chronic hepatic disease. e.g. chronic alcoholism. Wilson's disease.
4. Poorly controlled type I or type 2 diabetes mellitus
5. Donation or loss more than 400 ml blood within 60 days of baseline.
6. Known serious allergies to nucleoside/nucleotide analogs.
7. Subjects who are pregnant, nursing, or unwilling to use appropriate form of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Value of log10 hepatitis B virus (HBV) DNA decreases form baseline. | 48 weeks
Histological response | 48 weeks

SECONDARY OUTCOMES:
Percent of patients with hepatitis B virus (HBV) DNA below limit of detection (LOD) at week 48 with polymerase chain reaction (PCR) assay. | 48 weeks
Percent of patients with normalization of alanine aminotransferase (ALT) at week 48 | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, Principal Investigator — Xiangya Hospital
Locations (1):
- Xiangya hospital, Changsha, Hunan, China